CLINICAL TRIAL: NCT04001725
Title: Efficacy of metfOrmin in PrevenTIng Glucocorticoid-induced Diabetes in Melanoma, breAst or Lung Cancer Patients With Brain Metastases: the Phase II OPTIMAL Study
Brief Title: Efficacy of metfOrmin in PrevenTIng Glucocorticoid-induced Diabetes in Patients With Brain Metastases
Acronym: OPTIMAL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: University of Milan (Other)
Responsible Party: Principal Investigator, Filippo de Braud, Professor, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INT31/19; B43C17000350001 (Other Grant/Funding Number: Italian Minister of Health (5x1000 year 2014)); 2019-000105-73 (EudraCT Number)
Record Dates: First submitted 2019-06-04; First posted 2019-06-28 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Brain Metastases; Melanoma; Lung Cancer; Breast Cancer
Keywords: Metformin; Dexamethasone; Diabetes; Glucocorticoids; Phase II; Tumor; Immune system; Immunological Effects; Metabolic Effects; Anticancer Effects; Randomization; Quality of Life
MeSH Terms: conditions — Brain Neoplasms; Melanoma; Lung Neoplasms; Breast Neoplasms; Diabetes Mellitus; Neoplasms | interventions — Dexamethasone; Metformin

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized in a 1:1 ratio. Randomization will be stratified by means of minimization technique according to the following factors: primary tumor (melanoma versus lung versus breast cancer), dexamethasone dosage (8-12 mg vs >12 mg daily), baseline (pre-enrollment) fasting glycemia (< 100 versus 100-125 mg/dl). Patients randomized to the experimental arm will discontinue metformin after 30 days, unless diabetes has developed in the meanwhile and the physician believes that metformin is still required for its management. Patients randomized to the control arm who develop steroid-induced diabetes will be prescribed metformin, unless contraindicated, as the preferred therapy option for the management of hyperglycemia. In both treatment arms, dexamethasone will be administered until necessary and at the required dosage in the judgment of the treating physician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Dexamethasone) (Active Comparator): Patients subjected at a minimum daily dosage of 8 mg through the oral, intramuscular or intravenous administration route (control arm). The total dose can either administered once a day or through a refracted schedule
  Interventions: Drug: Dexamethasone
- B (Dexamethasone and Metformin) (Experimental): Patients subjected at a minimum daily dosage of 8 mg through the oral, intramuscular or intravenous administration route.The total dose can either administered once a day or through a refracted schedule.
  The same patients subjected at a metformin. Metformin initial dosage will be 850 mg per day, and will be escalated based on patient tolerability up to a maximum of 2550 mg daily (experimental arm).
  Interventions: Drug: Dexamethasone; Drug: Metformin

INTERVENTIONS:
Drug: Dexamethasone — A minimum daily dosage of 8 mg through the oral, intramuscular or intravenous administration route, once or twice a day.
Drug: Metformin — A minimum daily dosage of Dexamethasone 8 mg through the oral, intramuscular or intravenous administration route, once or twice a day and 2550 mg daily (maximum dose), oral administration (OS) of Metformin; starting dose will be 850 mg/day, to be progressively increased to 1700 mg/day on day 4 and 2550 mg/day on day 7, if well tolerated.
  Other Names: METFORAL
  Arms: B (Dexamethasone and Metformin)

SUMMARY:
This is a monocentric, open label, randomized Phase II study in patients with brain metastasis from melanoma, lung or breast cancer, who require treatment with high-dose dexamethasone, as defined as a minimum of 8 mg daily based on the clinician judgment, for at least three weeks, with or without radiation therapy. The aim is to investigate the metformin efficacy in preventing the onset of glucocorticoid-induced diabetes and other metabolic perturbations in patients with brain metastases from melanoma, lung or breast cancer.

DETAILED DESCRIPTION:
The study will be conducted in approximately 110 adult patients. aim of the study is to evaluate the effect of oral metformin in preventing GC-induced alterations of systemic metabolism, and in particular GC-induced diabetes. Other clinical objectives of the study consist in investigating the impact of metformin on precocious mortality, deterioration of ECOG PS and local (brain) disease control rate at one month. As an exploratory analysis, the effect of dexamethasone plus/minus metformin on other metabolites or growth factors (including amino acids, fatty acids, ketone bodies, IGF-1), as well as on the number, activation status and metabolism of peripheral blood immune cell populations will be evaluated

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 75 years
2. Histologically confirmed diagnosis of melanoma, lung (SCLC or NSCLC) or breast cancer
3. Recent (28 days), radiologically documented (contrast-enhanced CT or MRI) diagnosis of measurable brain metastases requiring treatment with high-dose dexamethasone (at least 8 mg daily for at least 21 days) plus/minus radiation therapy (RT).
4. Any previous or ongoing antitumor systemic therapy; patients who have never received previous systemic therapy can be also included.
5. Fasting glycemia < 126 mg/dl at the baseline evaluation or random glycemia of less than 200 mg/dl if the patient has not fasted for at least 8 hours before blood sampling.
6. Adequate blood tests:

   * Hemoglobin ≥ 9 g/dl
   * Absolute neutrophil count (ANC) in the range between 1.5-10 x 103/μl
   * Total bilirubin ≤ 1.5 times the upper normal limit (UNL). For patients with Gilbert syndrome or known liver metastases, bilirubin levels ≤ 3 times the UNL are considered acceptable
   * AST, ALT ≤ 3 times the UNL
   * Alkaline phosphatase ≤ 2.5 times the UNL
   * Serum creatinine concentration ≤ 1.5 x UNL
7. ECOG Performance Status ≤ 2
8. Life expectancy > 6 weeks
9. Written informed consent
10. Ability to swallow metformin tablets
11. Patients of female gender with the potential of childbearing (neither surgically sterile nor 2 years postmenopausal) must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for at least 60 days after study conclusion. Acceptable methods of contraception include double barrier method [i.e. condom and occlusive cap (diaphragm or cervical vault caps)] spermicide, intrauterine device (IUD), or steroidal contraceptive (oral, transdermal, implanted, or injected) in conjunction with a barrier method.
12. Patients of male gender having female partners with childbearing potential must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 60 days after participation in the study

Exclusion Criteria:

1. Leptomeningeal carcinomatosis, either radiologically documented or cytologically confirmed
2. History of brain metastases
3. Diagnosis of other malignancies in the last 5 years, except for superficial, radically treated basal cell carcinomas of the skin or in situ carcinomas of the cervix
4. Previous or current use of metformin
5. Ongoing therapy with systemic glucocorticoids at a dosage that is higher than 10 mg prednisone equivalent. Previous GC treatment is allowed if stopped at least 2 months before enrollment. Inhaled or topical steroids are permitted.
6. Diagnosis of Type 1 or Type 2 diabetes mellitus
7. Known history of HBV- or HCV-related infection
8. Known liver cirrhosis, even in the absence of significant alterations in blood tests
9. Clinically uncontrolled disorders of the lung, kidney, liver or cardio-vascular apparatus
10. Known history of HIV infection
11. Serious neurological or psychiatric disorders
12. Absence of a caregiver for patients with an ECOG performance status of 2
13. Pregnancy or lactation
14. Body mass index < 18.5 kg/m2
15. Past or current alcohol abuse (> 36 grams/day for men and 24grams/day for women)
16. Documented metabolic acidosis from any cause in the last 5 years
17. History of allergy or hypersensitivity to study drug components

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Metformin in preventing precocious (14 days) dexamethasone-induced diabetes | 14 days
  To evaluate the efficacy of metformin in preventing precocious (14 days) dexamethasone-induced diabetes, as defined as fasting plasma glucose levels ≥ 126 mg/dl, in patients with brain metastases from melanoma, lung or breast cancer.

SECONDARY OUTCOMES:
Dexamethasone-induced diabetes at 30 days | 30 days
  To study the efficacy of metformin in preventing dexamethasone-induced diabetes at 7 and 30 days after dexamethasone initiation, as defined as fasting plasma glucose levels ≥ 126 mg/dl, in patients with brain metastases from melanoma, lung or breast
Short-term mortality | 90 days
  To evaluate the efficacy of metformin in modifying short-term mortality (3 months) in patients taking high-dose dexamethasone
Brain local control rate of disease | 30 days
  To evaluate the efficacy of metformin in modifying the local disease control rate (brain) in patients treated with radiation therapy (RT) plus dexamethasone at 1 month
Patient ECOG performance status (PS) | 30 days
  To test the impact of metformin on precocious modifycation of patient ECOG Performance Status (PS) at 1 month after initiation of dexamethasone therapy.
Patient Quality of Life (QoL) | 30 days
  Patient QoL will be evaluated through the European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) C-30 version 3.0. The EORTC QLQ.C30 instrument will be scored according to the EORTC guidelines.
Absolute counts of immune cell populations | 2 years
  To investigate the potential impact of metformin on absolute counts of immune cell populations
Relative counts of immune cell populations | 2 years
  To investigate the potential impact of metformin on relative counts and activation status of activated antitumor lymphocytes
Activation status of immune cell populations | 2 years
  To investigate the potential impact of metformin on activated antitumor lymphocytes
Plasma lipids profile | 14 days
  To study the effect of metformin in modifying the plasma lipid profile at 14 days after treatment initiation
Plasma lipids profile | 30 days
  To study the effect of metformin in modifying the plasma lipid profile at 30 days after treatment initiation
Systemic inflammatory parameters | 2 years
  To investigate the effect of metformin on systemic plasma cytokines (G-CSF, GM-CSF, CCL2, VEGFA)
GC-induced changes in gut microbiota populations | 30 days
  To evaluate the impact of high-dose GCs on gut microbiota populations (30 days)
Metformin-induced changes in gut microbiota populations | 30 days
  To evaluate the impact of metformin on gut microbiota populations (30 days)
Amino acid profile | 14 days
  To study the effect of metformin in modifying the plasma amino acid profile at 14 days after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Filippo De Braud, Professor, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanahan D, Weinberg RA. Hallmarks of cancer: the next generation. Cell. 2011 Mar 4;144(5):646-74. doi: 10.1016/j.cell.2011.02.013. PMID 21376230
- [Background] Vernieri C, Casola S, Foiani M, Pietrantonio F, de Braud F, Longo V. Targeting Cancer Metabolism: Dietary and Pharmacologic Interventions. Cancer Discov. 2016 Dec;6(12):1315-1333. doi: 10.1158/2159-8290.CD-16-0615. Epub 2016 Nov 21. PMID 27872127
- [Background] O'Neill LA, Kishton RJ, Rathmell J. A guide to immunometabolism for immunologists. Nat Rev Immunol. 2016 Sep;16(9):553-65. doi: 10.1038/nri.2016.70. Epub 2016 Jul 11. PMID 27396447
- [Background] Lin X, DeAngelis LM. Treatment of Brain Metastases. J Clin Oncol. 2015 Oct 20;33(30):3475-84. doi: 10.1200/JCO.2015.60.9503. Epub 2015 Aug 17. PMID 26282648
- [Background] Harris D, Barts A, Connors J, Dahl M, Elliott T, Kong J, Keane T, Thompson D, Stafford S, Ur E, Sirrs S. Glucocorticoid-induced hyperglycemia is prevalent and unpredictable for patients undergoing cancer therapy: an observational cohort study. Curr Oncol. 2013 Dec;20(6):e532-8. doi: 10.3747/co.20.1499. PMID 24311953
- [Background] Weiser MA, Cabanillas ME, Konopleva M, Thomas DA, Pierce SA, Escalante CP, Kantarjian HM, O'Brien SM. Relation between the duration of remission and hyperglycemia during induction chemotherapy for acute lymphocytic leukemia with a hyperfractionated cyclophosphamide, vincristine, doxorubicin, and dexamethasone/methotrexate-cytarabine regimen. Cancer. 2004 Mar 15;100(6):1179-85. doi: 10.1002/cncr.20071. PMID 15022284
- [Background] Furnary AP, Gao G, Grunkemeier GL, Wu Y, Zerr KJ, Bookin SO, Floten HS, Starr A. Continuous insulin infusion reduces mortality in patients with diabetes undergoing coronary artery bypass grafting. J Thorac Cardiovasc Surg. 2003 May;125(5):1007-21. doi: 10.1067/mtc.2003.181. PMID 12771873
- [Background] Perez A, Jansen-Chaparro S, Saigi I, Bernal-Lopez MR, Minambres I, Gomez-Huelgas R. Glucocorticoid-induced hyperglycemia. J Diabetes. 2014 Jan;6(1):9-20. doi: 10.1111/1753-0407.12090. Epub 2013 Oct 29. PMID 24103089
- [Background] Oyer DS, Shah A, Bettenhausen S. How to manage steroid diabetes in the patient with cancer. J Support Oncol. 2006 Oct;4(9):479-83. No abstract available. PMID 17080737
- [Background] Bozzi F, Mogavero A, Varinelli L, Belfiore A, Manenti G, Caccia C, Volpi CC, Beznoussenko GV, Milione M, Leoni V, Gloghini A, Mironov AA, Leo E, Pilotti S, Pierotti MA, Bongarzone I, Gariboldi M. MIF/CD74 axis is a target for novel therapies in colon carcinomatosis. J Exp Clin Cancer Res. 2017 Jan 23;36(1):16. doi: 10.1186/s13046-016-0475-z. PMID 28114961
- [Background] Wallace MD, Metzger NL. Optimizing the Treatment of Steroid-Induced Hyperglycemia. Ann Pharmacother. 2018 Jan;52(1):86-90. doi: 10.1177/1060028017728297. Epub 2017 Aug 24. PMID 28836444
- [Background] Kwon S, Hermayer KL, Hermayer K. Glucocorticoid-induced hyperglycemia. Am J Med Sci. 2013 Apr;345(4):274-277. doi: 10.1097/MAJ.0b013e31828a6a01. PMID 23531958
- [Background] Zhang ZJ, Bi Y, Li S, Zhang Q, Zhao G, Guo Y, Song Q. Reduced risk of lung cancer with metformin therapy in diabetic patients: a systematic review and meta-analysis. Am J Epidemiol. 2014 Jul 1;180(1):11-4. doi: 10.1093/aje/kwu124. Epub 2014 Jun 10. PMID 24920786
- [Background] Bodmer M, Meier C, Krahenbuhl S, Jick SS, Meier CR. Long-term metformin use is associated with decreased risk of breast cancer. Diabetes Care. 2010 Jun;33(6):1304-8. doi: 10.2337/dc09-1791. Epub 2010 Mar 18. PMID 20299480
- [Background] Pusceddu S, Vernieri C, Di Maio M, Marconcini R, Spada F, Massironi S, Ibrahim T, Brizzi MP, Campana D, Faggiano A, Giuffrida D, Rinzivillo M, Cingarlini S, Aroldi F, Antonuzzo L, Berardi R, Catena L, De Divitiis C, Ermacora P, Perfetti V, Fontana A, Razzore P, Carnaghi C, Davi MV, Cauchi C, Duro M, Ricci S, Fazio N, Cavalcoli F, Bongiovanni A, La Salvia A, Brighi N, Colao A, Puliafito I, Panzuto F, Ortolani S, Zaniboni A, Di Costanzo F, Torniai M, Bajetta E, Tafuto S, Garattini SK, Femia D, Prinzi N, Concas L, Lo Russo G, Milione M, Giacomelli L, Buzzoni R, Delle Fave G, Mazzaferro V, de Braud F. Metformin Use Is Associated With Longer Progression-Free Survival of Patients With Diabetes and Pancreatic Neuroendocrine Tumors Receiving Everolimus and/or Somatostatin Analogues. Gastroenterology. 2018 Aug;155(2):479-489.e7. doi: 10.1053/j.gastro.2018.04.010. Epub 2018 Apr 13. PMID 29655834
- [Background] Seelig E, Meyer S, Timper K, Nigro N, Bally M, Pernicova I, Schuetz P, Muller B, Korbonits M, Christ-Crain M. Metformin prevents metabolic side effects during systemic glucocorticoid treatment. Eur J Endocrinol. 2017 Mar;176(3):349-358. doi: 10.1530/EJE-16-0653. Epub 2017 Jan 10. PMID 28073907
- [Background] Bostrom B, Uppal P, Chu J, Messinger Y, Gandrud L, McEvoy R. Safety and efficacy of metformin for therapy-induced hyperglycemia in children with acute lymphoblastic leukemia. J Pediatr Hematol Oncol. 2013 Oct;35(7):504-8. doi: 10.1097/MPH.0b013e31829cdeba. PMID 23823111
- [Derived] Green BJ, Marazzini M, Hershey B, Fardin A, Li Q, Wang Z, Giangreco G, Pisati F, Marchesi S, Disanza A, Frittoli E, Martini E, Magni S, Beznoussenko GV, Vernieri C, Lobefaro R, Parazzoli D, Maiuri P, Havas K, Labib M, Sigismund S, Fiore PPD, Gunby RH, Kelley SO, Scita G. PillarX: A Microfluidic Device to Profile Circulating Tumor Cell Clusters Based on Geometry, Deformability, and Epithelial State. Small. 2022 Apr;18(17):e2106097. doi: 10.1002/smll.202106097. Epub 2022 Mar 28. PMID 35344274